CLINICAL TRIAL: NCT04812678
Title: Interest of DBM Fasciatherapy for Physiotherapy in the Care of Patients Suffering From Non-Specific Chronic Low Back Pain: a Cluster Randomized Multicenter Clinical Trial
Brief Title: Efficacy of DBM Fasciatherapy for Patients Suffering From Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FasciaFrance (Other)
Collaborators: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF2021
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; DBM Fasciatherapy; Physiotherapy; Manual Therapy; Fascia
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapy (Active Comparator): Conventional physiotherapy, in line with french "Haute Autorité de Santé" guidelines
  Interventions: Procedure: Physiotherapy
- Physiotherapy and Fasciatherapy (Experimental): Conventional physiotherapy, in line with french "Haute Autorité de Santé" guidelines, associated with Fasciatherapy Danis Bois Method
  Interventions: Procedure: Fasciatherapy; Procedure: Physiotherapy
- Fasciatherapy (Experimental): Fasciatherapy Danis Bois Method
  Interventions: Procedure: Fasciatherapy

INTERVENTIONS:
Procedure: Fasciatherapy — Fasciatherapy, with manual therapy and/or gestual therapy.
  Other Names: DBM Fasciatherapy; Danis Bois Method Fasciatherapy
  Arms: Fasciatherapy; Physiotherapy and Fasciatherapy
Procedure: Physiotherapy — Conventional physiotherapy with massage, exercises, electrotherapy, vertebral traction, heat, cold.
  Other Names: Physical Therapy
  Arms: Physiotherapy; Physiotherapy and Fasciatherapy

SUMMARY:
Low back pain (LBP) is pain localized below the costal margin and above the inferior gluteal folds. It may be associated with radiculalgia. Non-specific LBP refers to LBP without specific problems such as infection, inflammation, vertebral fracture or cancer. Chronic LBP is a LBP lasting more than 3 months.

The causes of LBP remain unknown. While there are recommendations for physiotherapy, the protocol of care is not well defined. New therapeutic models centered on neurophysiology are replacing biomechanics-based models. New programs centered on patient education and a biopsychosocial approach are emerging.

Research has shown the possible involvement of fascia in LBP and the interest of manual fascia therapies in the treatment of LBP. To date, there are no studies that have shown the effects of fasciatherapy in the treatment of non-specific LBP.

In France, many physiotherapists use this type of treatment and more specifically fasciatherapy. French physiotherapists say that it may improve their management of LBP. Studies on fasciatherapy have highlighted the effects of fasciatherapy in the management of fibromyalgia pain, the treatment of anxiety, malaise and the improvement of body perception. They show the multidimensional actions of fasciatherapy and support its clinical, functional and psychosocial evaluation for LBP.

Fasciatherapy is part of the manual therapies that target their action on the fascial system. This "patient-centered" technique is a biopsychosocial and humanistic approach to health. The manual and gestural approaches of the fascia are part of the Non-Pharmaceutical Interventions field. Fasciatherapy involves manual and gestural interventions, with the objective of restoring the contractile, elastic and movement properties of the fascia in order to provide relief, improve function and quality of life for patients.

In France, fasciatherapy is not part of recommendations and is not recognized by the Conseil National de l'Ordre des Masseurs-Kinésithérapeutes.

This study aims to assess the effects of fasciatherapy on LBP and to evaluate how it could contribute to its management for physiotherapists. It is a cluster randomized trial conducted on 180 subjects. Intensity of pain (measured with VAS) is the primary outcome. The secondary outcomes are the impact of LBP on daily life (Dallas Pain Questionnaire), on quality of life (SF-12 questionnaire), on anxiety (STAI questionnaire), and the evolution of drug consumption.

The study will take place in France and the treatment structures will be the practitioners' practice.

ELIGIBILITY:
Inclusion Criteria:

* First consultation for Low Back Pain with the practitioner
* Having a diagnostic of chronic non-specific Low Back Pain based on the French Haute Autorité de Santé guidelines (https://www.has-sante.fr/upload/docs/application/pdf/2019-04/fm_lombalgie_v2_2.pdf):
* excluding specific Low Back Pain (tumor, infection, inflammation, etc.)
* no red flag
* Low Back Pain for more than 3 months
* Having had the French validated version of:
* evaluation of pain intensity with Visual Analog Scale
* STarT Back Screening Tool questionnaire
* Dallas Pain questionnaire

Exclusion Criteria:

* Specific Low Back Pain (rheumatologist disease, tumoral compression, central neurological pathology, etc.)
* Psychiatric disorder (apart from the usual co-morbidities of chronic low back pain)
* Pregnancy or breastfeeding
* Being under guardianship or curatorship
* Deprivation of liberty or legal protection measure
* Being unable to give consent
* Being unable of fill out a questionnaire

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Courraud, PhD, PT, Study Director — Centre d'Etude et de Recherche Appliquée en Psychopédagogie perceptive - University Fernando Pessoa
Locations (1):
- FasciaFrance, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Background] Bruyere O, Demoulin M, Beaudart C, Hill JC, Maquet D, Genevay S, Mahieu G, Reginster JY, Crielaard JM, Demoulin C. Validity and reliability of the French version of the STarT Back screening tool for patients with low back pain. Spine (Phila Pa 1976). 2014 Jan 15;39(2):E123-8. doi: 10.1097/BRS.0000000000000062. PMID 24108286
- [Background] Marty M, Blotman F, Avouac B, Rozenberg S, Valat JP. Validation of the French version of the Dallas Pain Questionnaire in chronic low back pain patients. Rev Rhum Engl Ed. 1998 Feb;65(2):126-34. PMID 9540121
- [Background] Leplege A, Ecosse E, Verdier A, Perneger TV. The French SF-36 Health Survey: translation, cultural adaptation and preliminary psychometric evaluation. J Clin Epidemiol. 1998 Nov;51(11):1013-23. doi: 10.1016/s0895-4356(98)00093-6. PMID 9817119
- [Background] Lawlis GF, Cuencas R, Selby D, McCoy CE. The development of the Dallas Pain Questionnaire. An assessment of the impact of spinal pain on behavior. Spine (Phila Pa 1976). 1989 May;14(5):511-6. doi: 10.1097/00007632-198905000-00007. PMID 2524890
- [Background] Ware J, Kolinski M, Keller S. How to score the SF-12 physical and mental health summaries: a user's manual. Boston: The Health Institute, New England Medical Centre, Boston, MA. 1995;
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Boureau F. L'appréciation de la sévérité d'une douleur chronique. Médecine et hygiène. 1987;45(1703):1560-6.
- [Background] Wilke J, Schleip R, Klingler W, Stecco C. The Lumbodorsal Fascia as a Potential Source of Low Back Pain: A Narrative Review. Biomed Res Int. 2017;2017:5349620. doi: 10.1155/2017/5349620. Epub 2017 May 11. PMID 28584816
- [Background] Courraud C, Bois D, Lieutaud A. Apports de la pratique de la fasciathérapie à l'exercice de la physiothérapie: le point de vue des praticiens. Mains Libres. 2016;(3):49-58.
- See also: French Haute Autorité de Santé guidelines for the treatment of non-specific Low Back Pain — https://www.has-sante.fr/upload/docs/application/pdf/2019-04/fm_lombalgie_v2_2.pdf

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Physiotherapy/fasciatherapy practices
Groups:
- Active Comparator: Physiotherapy: Procedure: Physiotherapy Conventional physiotherapy with massage, exercises, electrotherapy, vertebral traction, heat, cold.
  Other Names:
  Physical Therapy
- Experimental: Physiotherapy and Fasciatherapy: Procedure: Fasciatherapy Fasciatherapy, with manual therapy and/or gestual therapy.
  Other Names:
  DBM Fasciatherapy Danis Bois Method Fasciatherapy Procedure: Physiotherapy Conventional physiotherapy with massage, exercises, electrotherapy, vertebral traction, heat, cold.
  Other Names:
  Physical Therapy
- Experimental: Fasciatherapy: Procedure: Fasciatherapy Fasciatherapy, with manual therapy and/or gestual therapy.
  Other Names:
  DBM Fasciatherapy Danis Bois Method Fasciatherapy
Period: Overall Study
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Started | 63; 20 Physiotherapy/fasciatherapy practices | 62; 20 Physiotherapy/fasciatherapy practices | 63; 20 Physiotherapy/fasciatherapy practices
Completed | 63; 20 Physiotherapy/fasciatherapy practices | 62; 20 Physiotherapy/fasciatherapy practices | 63; 20 Physiotherapy/fasciatherapy practices
Not Completed | 0; 0 Physiotherapy/fasciatherapy practices | 0; 0 Physiotherapy/fasciatherapy practices | 0; 0 Physiotherapy/fasciatherapy practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy | Total
Number analyzed (Participants) | 63 | 62 | 63 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (7.9) | 45.8 (7.7) | 47.6 (7.1) | 46.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 38 | 124
  Male | 22 | 17 | 25 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Star Back outil Triant [Mean (Standard Deviation); unit: units on a scale] — five questions: 1. fear, 2. anxiety, 3. catastrophizing, 4. feeling depressed, and 5. embarrassment.
  four questions on physical risk factors for poorer prognosis: 1. referred leg pain, 2. neck/shoulder pain, 3. inability to walk, and 4. difficulty dressing.
  The overall score ranges from 0 to 9 (best to worst), and divides the population into groups with a low, medium and high risk of a poorer prognosis.
  global score ≤3, low prognostic risk. combined global score ≥4, medium prognostic risk global score ≥7, high-risk category.
  units on a scale | 4.35 (1.93) | 4.63 (2.09) | 3.94 (1.91) | 4.3 (1.98)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Before the 1st session (start of the study for the patient)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 4.2 (2.4) | 4.1 (2.2) | 4.0 (2.1)

2. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: After the 1st session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 2.9 (2.3) | 2.9 (2.2) | 2.6 (2.1)

3. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Before the 2nd session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 3.7 (2.2) | 3.7 (2.6) | 3.1 (2.4)

4. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: After the 2nd session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 2.3 (1.8) | 2.3 (2.1) | 2.2 (2.0)

5. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Before the 3rd session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 3.1 (2.2) | 3.4 (2.3) | 2.9 (2.3)

6. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: After the 3rd session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 2.0 (1.9) | 2.1 (2.1) | 1.7 (1.8)

7. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Before the 4th session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 2.9 (2.3) | 2.5 (2.0) | 2.2 (1.9)

8. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: After the 4th session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 1.9 (1.9) | 1.8 (1.8) | 1.5 (1.6)

9. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Before the 5th session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 3.0 (2.5) | 2.2 (1.9) | 2.1 (2.1)

10. Primary Outcome: Pain Intensity
Description: Measure of pain intensity with Visual Analog Scale: 0 (no pain) to 10 (worst imaginable pain)
Time Frame: After the 5th session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 1.8 (1.9) | 1.4 (1.5) | 1.4 (1.7)

11. Secondary Outcome: Change in Trait of Anxiety
Description: Evaluation of the change in trait of anxiety with State Trait Inventory Anxiety questionnaire, part Y-B: scale from 20 (no anxiety) to 80 (maximum anxiety)
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 61 | 62 | 63
units on a scale | 40.3 (9.7) | 45.0 (9.5) | 43.0 (11.0)

12. Secondary Outcome: Evaluation of State of Anxiety
Description: Evaluation of the change in state of anxiety with State Trait Inventory Anxiety questionnaire, part Y-A: scale from 20 (no anxiety) to 80 (maximum anxiety)
Time Frame: Before the 1st session (start of the study for the patient)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 36.9 (9.5) | 42.1 (11.6) | 41.8 (13.1)

13. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: After the 1st session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 28.0 (6.2) | 30.0 (6.6) | 30.2 (8.5)

14. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: Before the 2nd session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 34.2 (9.0) | 40.2 (11.7) | 35.5 (11.8)

15. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: After the 2nd session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 28.3 (6.8) | 31.6 (7.9) | 29.0 (9.1)

16. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: Before the 3rd session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 32.6 (8.1) | 38.8 (11.6) | 36.0 (12.4)

17. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: After the 3rd session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 27.3 (6.7) | 31.0 (8.5) | 28.8 (9.4)

18. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: Before the 4th session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 34.2 (9.6) | 36.6 (13.2) | 34.9 (11.8)

19. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: After the 4th session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 28.8 (7.7) | 30.4 (9.8) | 29.0 (9.3)

20. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: Before the 5th session (within a total timeframe of 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 34.5 (10.9) | 35.9 (11.9) | 35.3 (12.1)

21. Secondary Outcome: Evaluation of State of Anxiety
Description: as for outcome 12
Time Frame: After the 5th session (30 to 45 minutes after the previous measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 28.9 (8.4) | 29.4 (8.5) | 28.8 (10.1)

22. Secondary Outcome: Analgesic Consumption
Description: Evaluation of analgesic consumption (interview of the patient)
Time Frame: 1st session (start of the study for the patient)
Measure: Number; unit: participants
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
participants | 14 | 10 | 21

23. Secondary Outcome: Analgesic Consumption
Description: Evaluation of analgesic consumption (interview of the patient)
Time Frame: 2nd session (within a total timeframe of 3 months)
Measure: Number; unit: participants
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
participants | 9 | 13 | 18

24. Secondary Outcome: Analgesic Consumption
Description: Evaluation of analgesic consumption (interview of the patient)
Time Frame: 3rd session (within a total timeframe of 3 months)
Measure: Number; unit: participants
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
participants | 15 | 9 | 17

25. Secondary Outcome: Analgesic Consumption
Description: Evaluation of analgesic consumption (interview of the patient)
Time Frame: 4th session (within a total timeframe of 3 months)
Measure: Number; unit: participants
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
participants | 13 | 14 | 9

26. Secondary Outcome: Analgesic Consumption
Description: Evaluation of analgesic consumption (interview of the patient)
Time Frame: 5th session (within a total timeframe of 3 months)
Measure: Number; unit: participants
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
participants | 13 | 7 | 8

27. Secondary Outcome: Change in Trait of Anxiety
Description: as for outcome 11
Time Frame: After the last (5st) session, in a timeframe of 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
units on a scale | 38.9 (11.0) | 42.0 (11.2) | 40.2 (11.7)

28. Secondary Outcome: Change in the Quality of Life - Physical Score
Description: Assessment of the change in the quality of life with the French version of the short version (SF-12) of "Short Form with 36 questions" (SF-36) questionnaire: scale from 0 (bad) to 100 (best)
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 62 | 61 | 63
score on a scale | 39.8 (7.0) | 40.5 (8.7) | 41.6 (8.3)

29. Secondary Outcome: Change in the Quality of Life - Physical Score
Description: as for outcome 28
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 61 | 60 | 61
score on a scale | 42.4 (8.5) | 46.1 (8.6) | 46.7 (8.3)

30. Secondary Outcome: Change in the Quality of Life - Mental Score
Description: as for outcome 28
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 62 | 61 | 63
score on a scale | 45.9 (9.5) | 40.3 (10.0) | 44.7 (9.5)

31. Secondary Outcome: Change in the Quality of Life - Mental Score
Description: as for outcome 28
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
Number analyzed (Participants) | 61 | 60 | 61
score on a scale | 47.7 (8.2) | 45.9 (9.9) | 47.2 (8.4)

32. Secondary Outcome: Change in Functional Abilities - Daily Activities
Description: Evaluation of the functional disability change, with French version of Dallas Pain Questionnaire: 4 items evaluated from 0 (no impact) to 100% (maximun impact)
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 62
score on a scale | 54.0 (16.6) | 50.2 (18.2) | 49.4 (18.2)

33. Secondary Outcome: Change in Functional Abilities - Daily Activities
Description: as for outcome 32
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 40.1 (19.3) | 32.5 (20.1) | 30.8 (19.7)

34. Secondary Outcome: Change in Functional Abilities - Professional and Leisure Activities
Description: as for outcome 32
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 60 | 63
score on a scale | 44.2 (20.4) | 44.1 (20.8) | 43.8 (23.2)

35. Secondary Outcome: Change in Functional Abilities - Professional and Leisure Activities
Description: as for outcome 32
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 61 | 60
score on a scale | 33.8 (21.9) | 25.5 (21.7) | 28.6 (24.3)

36. Secondary Outcome: Change in Functional Abilities - Anxiety and Depression
Description: as for outcome 32
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 61 | 62
score on a scale | 32.1 (19.7) | 35.1 (18.6) | 32.7 (23.0)

37. Secondary Outcome: Change in Functional Abilities - Anxiety and Depression
Description: as for outcome 32
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 61 | 60
score on a scale | 27.5 (24.1) | 26.1 (21.9) | 25.2 (21.2)

38. Secondary Outcome: Change in Functional Abilities - Sociability
Description: as for outcome 32
Time Frame: Before the 1st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 63
score on a scale | 23.1 (19.8) | 24.4 (20.3) | 23.6 (21.4)

39. Secondary Outcome: Change in Functional Abilities - Sociability
Description: as for outcome 32
Time Frame: After the 5st session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy | Physiotherapy and Fasciatherapy | Fasciatherapy
Number analyzed (Participants) | 63 | 62 | 61
score on a scale | 18.0 (16.4) | 19.3 (19.8) | 16.7 (19.7)

ADVERSE EVENTS:
Time Frame: 16 months
Description: There was no risk
Arm/Group | Active Comparator: Physiotherapy | Experimental: Physiotherapy and Fasciatherapy | Experimental: Fasciatherapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/62 | 0/63

LIMITATIONS AND CAVEATS:
This study confirms the need to develop clinical research into fascia therapies for musculoskeletal disorders. A study could be carried out to verify the durability of the effects obtained, with assessments at 6 months and 1 year. Another study could be carried out using the same criteria and in comparison with other fascia therapies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT04812678/Prot_SAP_000.pdf